CLINICAL TRIAL: NCT01785602
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study Evaluating Efficacy and Safety of QAW039 in the Treatment of Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety Study of QAW039 in the Treatment of Patients With Moderate to Severe Atopic Dermatitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039X2201; 2012-005321-78 (EudraCT Number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic eczema; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- QAW039 (Experimental): Participants received QAW039 450 mg daily by mouth.
  Interventions: Drug: QAW039
- Placebo (Placebo Comparator): Participants received matching placebo to QAW039.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 — Capsules
  Arms: QAW039
Drug: Placebo — Capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether QAW039 is safe and has beneficial effects in people who have moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Key Inclusion Criteria:

* Presence of atopic dermatitis confirmed by Itchy skin condition in the past 12 months plus three, or more, of the following:

  * History of involvement of the skin creases (fronts of elbows, behind knees, fronts of ankles, around neck or around eyes)
  * Personal history of asthma or hay fever
  * History of generally dry skin in the past year
  * Onset before age of 2 years
  * Visible flexural dermatitis
* Patients with an EASI score of ≥15 at screening and stable AD (not currently experiencing an acute flare of their AD).
* Patients that have been treated with topical corticosteroids or topical calcineurin inhibitors on at least one occasion, or could not use topical drugs (due to contraindications, side effects, etc.) and are candidates for or have previously received systemic treatment.

Key Exclusion Criteria:

* History of hypersensitivity to any of the study drugs (including local anesthesia) or to drugs of similar chemical classes (CRTh2 antagonists)
* History of serious allergic reactions to any allergen, such as anaphylactic shock or life-threatening asthma, prior intubation, respiratory arrest, hospitalization due to asthma within the last 3 months or seizures as a result of asthma
* History of clinically significant ECG abnormalities or screening/baseline ECG that demonstrated clinical significant abnormalities which could affect patient safety or interpretation of study results
* History of long QT syndrome or whose QTc interval (Frederica's) was prolonged (>450 msec for males and females) at screening
* Use of topical prescription treatment (e.g., topical corticosteroids, calcineurin inhibitors, antibiotics, etc.) within two weeks prior to initial dosing of study drug. Patient use of emollients was encouraged
* Exception: For local atopic dermatitis flares during this 2-week interval, mild topical corticosteroids may be taken short term (up to one week)
* Recent previous systemic treatment with phototherapy, systemic antihistamines, immunosuppressive agents (e.g., cyclosporine, mycophenolate, or oral tacrolimus, including therapeutic proteins)
* Patients on maintenance immunotherapy who either began their allergen specific immunotherapy regimen or had a clinically relevant change to their immunotherapy within one month prior to granting informed consent
* Patients on high-dose statin therapy (>40 mg fluvastatin or 20 mg simvastatin, atorvastin, pravastatin, or rosuvastatin [10 mg if Asian])
* Excessive exposure to UV light in the three weeks prior to study start (screening), including tanning and sun beds and/or planning excessive sunbathing or beach holidays with associated sun bathing during the treatment period
* History of hypertrophic scarring
* Body mass index <17 or >40 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Australia (3):
  - Novartis Investigative Site, Phillip, Australian Capital Territory
  - Novartis Investigative Site, Benowa, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
- Novartis Investigative Site, Vienna, Austria
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Novartis Investigative Site, Sofia, Bulgaria, Bulgaria
- Germany (4):
  - Novartis Investigative Site, Dresden, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Münster
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Durban, South Africa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QAW039 | Placebo
Started | 76 | 27
Completed | 63 | 18
Not Completed | 13 | 9
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 3 | 5
Not completed — Administrative problems | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 | Placebo | Total
Number analyzed (Participants) | 76 | 27 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.5 (13.08) | 38.7 (9.95) | 36.3 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 12 | 39
  Male | 49 | 15 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI)
Description: Investigators assessed presence and severity of erythema, induration/papulation, excoriation, and lichenification in four body areas: head/neck (H), upper limbs (UL), trunk (T), and lower limbs (LL). Investigators assigned a severity score from 0 - 3 for each area (none=0, mild=1, moderate=2, and severe=3). Investigators could assign half-points. Investigators also assigned an area score from 0 (no atopic dermatitis lesion in the area) to 6 (entire area is affected) for each area. The weighting factor was 0.1 for head/neck, 0.2 for upper limbs, 0.3 for trunk, and 0.4 for lower limbs. The total body score for each body region was obtained by multiplying the sum of the severity scores of the four key signs by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gave the EASI total, ranging from 0 to 72. A higher score represented greater disease severity. A negative change from baseline indicates improvement.
Time Frame: Baseline, 12 weeks
Population: All randomized participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 76 | 27
Score on a scale | -8.65 (0.010) | -6.95 (0.017)

2. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index
Description: as for outcome 1
Time Frame: Baseline, 4 weeks, 8 weeks
Population: All randomized participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 76 | 27
Score on a scale
  Week 4 | -6.22 (0.010) | -5.89 (0.017)
  Week 8 | -7.49 (0.010) | -5.61 (0.017)

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from day 1 until 4 weeks after end of study (week 20)
Arm/Group | QAW039 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/76 | 4/27
Other Adverse Events (participants affected / at risk) | 44/76 | 16/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 (N=76) | Placebo (N=27)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 (N=76) | Placebo (N=27)
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 2
Nausea (Gastrointestinal disorders) | 6 | 3
Fatigue (General disorders) | 5 | 1
Nasopharyngitis (Infections and infestations) | 11 | 1
Oral herpes (Infections and infestations) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 7 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 2
Tension headache (Nervous system disorders) | 1 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 24 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Hot flush (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.